CLINICAL TRIAL: NCT05864586
Title: Nicotine Concentration and Forms: Differential Appeal to Smokers Versus Non-Smokers
Brief Title: Developing E-liquid Product Standards (Sweet Spot Study)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Responsible Party: Principal Investigator, Theodore Wagener, Principal Investigator, Ohio State University Comprehensive Cancer Center
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Prevention
Other Study IDs: OSU-22253; NCI-2023-03206 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2023-05-09; First posted 2023-05-18 (Actual); Results first posted 2025-04-10 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-03

CONDITIONS: Nicotine; Nicotine Vaping; E-cigarette Use
MeSH Terms: conditions — Vaping

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Young adult EC users (Active Comparator): Young Adult EC users
  Interventions: Behavioral: Vaping study EC A; Behavioral: Vaping study EC B; Behavioral: Vaping study EC C; Behavioral: Vaping study EC D; Behavioral: Vaping study EC E; Behavioral: Vaping study EC F; Behavioral: Vaping study EC G; Behavioral: Vaping study EC H; Behavioral: Vaping study EC I; Behavioral: Vaping study EC J
- Older adult smokers (Active Comparator): Adult smokers
  Interventions: Behavioral: Vaping study EC A; Behavioral: Vaping study EC B; Behavioral: Vaping study EC C; Behavioral: Vaping study EC D; Behavioral: Vaping study EC E; Behavioral: Vaping study EC F; Behavioral: Vaping study EC G; Behavioral: Vaping study EC H; Behavioral: Vaping study EC I; Behavioral: Vaping study EC J

INTERVENTIONS:
Behavioral: Vaping study EC A — Vaping two puffs using the study EC device
Behavioral: Vaping study EC B — Vaping two puffs using the study EC device
Behavioral: Vaping study EC C — Vaping two puffs using the study EC device
Behavioral: Vaping study EC D — Vaping two puffs using the study EC device
Behavioral: Vaping study EC E — Vaping two puffs using the study EC device
Behavioral: Vaping study EC F — Vaping two puffs using the study EC device
Behavioral: Vaping study EC G — Vaping two puffs using the study EC device
Behavioral: Vaping study EC H — Vaping two puffs using the study EC device
Behavioral: Vaping study EC I — Vaping two puffs using the study EC device
Behavioral: Vaping study EC J — Vaping two puffs using the study EC device

SUMMARY:
The Sweet Spot Study aims to evaluate the effect of e-liquids with nicotine varying in freebase (FB) levels and concentrations on the appeal of electronic cigarettes (ECs) in young adult EC users with minimal/no history of smoking and older adult smokers.

ELIGIBILITY:
Inclusion criteria:

1. Young adult e-cigarette user or older adult smoker
2. Willing to abstain from all nicotine product use for 12 hours prior to the study visit
3. Read and speak English

Exclusion criteria:

1. Currently attempting to quit nicotine products
2. Currently pregnant, planning to become pregnant, or breastfeeding
3. Current or past use of tobacco products other than e-cigarettes or cigarettes
4. Self-reported diagnosis of lung disease
5. Self-reported new or unstable cardiovascular disease

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 150 (Actual)
Dates: Start 2023-05-30 (Actual); Primary Completion 2024-02-26 (Actual); Study Completion 2024-02-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Theodore L Wagener, PhD, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (1):
- Ohio State University Comprehensive Cancer Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cho YJ, Brinkman MC, Hinton A, Nshimiyimana JD, Mehta T, Adeniji A, Norton K, El Hellani A, Wagener TL. The sweet spot study-Developing e-liquid product standards for nicotine form and concentration to improve public health: Protocol for a randomized, double-blinded, crossover study. PLoS One. 2023 Sep 12;18(9):e0291522. doi: 10.1371/journal.pone.0291522. eCollection 2023. PMID 37699050
- See also: The Jamesline — http://cancer.osu.edu

RESULTS

PARTICIPANT FLOW:
Groups:
- Young Adult EC Users; Older Adult Smokers: Guided by study staff, young adult e-cigarette users and older adult smokers took two puffs from each of the 10 study conditions ([5%, 25%, 45%, 65%, 85%] freebase nicotine fractions × [20 mg/mL, 50 mg/mL] nicotine concentrations) using the study e-cigarette device. Each condition was administered in a single vaping session, with a 10-minute washout period between conditions. Participants received pre-filled e-liquid pods in random order and were instructed to inhale each puff for at least one second.
Period: Overall Study
Arm/Group | Young Adult EC Users | Older Adult Smokers
Started | 70 | 80
20mg/mL Nicotine Concentration, 5% Free-base Fraction Study EC Device | 66 | 67
20mg/mL Nicotine Concentration, 25% Free-base Fraction Study EC Device | 66 | 66
20mg/mL Nicotine Concentration, 45% Free-base Fraction Study EC Device | 66 | 66
20mg/mL Nicotine Concentration, 65% Free-base Fraction Study EC Device | 66 | 66
20mg/mL Nicotine Concentration, 85% Free-base Fraction Study EC Device | 66 | 67
50mg/mL Nicotine Concentration, 5% Free-base Fraction Study EC Device | 66 | 66
50mg/mL Nicotine Concentration, 25% Free-base Fraction Study EC Device | 66 | 66
50mg/mL Nicotine Concentration, 45% Free-base Fraction Study EC Device | 66 | 66
50mg/mL Nicotine Concentration, 65% Free-base Fraction Study EC Device | 66 | 66
50mg/mL Nicotine Concentration, 85% Free-base Fraction Study EC Device | 66 | 66
Completed | 66 | 66
Not Completed | 4 | 14
Not completed — Ineligible | 4 | 12
Not completed — Pregnancy | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Young Adult EC Users: Young adult e-cigarette users
- Older Adult Smokers: Older adult cigarette smokers
- Total: Total of all reporting groups
Arm/Group | Young Adult EC Users | Older Adult Smokers | Total
Number analyzed (Participants) | 66 | 67 | 133
Age, Continuous [Mean (Standard Deviation); unit: years] | 22.12 (1.16) | 39.39 (6.71) | 30.82 (9.91)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 51 | 53 | 104
  Male | 15 | 14 | 29
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 1 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 9 | 12
  White | 55 | 54 | 109
  More than one race | 4 | 3 | 7
  Unknown or Not Reported | 1 | 0 | 1
Cigarettes Smoked per Day [Mean (Standard Deviation); unit: cigarettes per day] | 0.02 (0.12) | 13.19 (6.33) | 6.65 (7.99)

OUTCOME MEASURES:

1. Primary Outcome: Behavioral Intentions for Continued Use
Description: Self-report measure on a 7-point scale completed following e-cigarette self-administration. Ratings range from1 (extremely unlikely) to 7 (extremely likely) with higher scores indicating a higher likelihood of continuing to use the product.
Time Frame: The outcome measure was assessed immediately after each vaping session. During each vaping session, participants took two puffs of each of the 10 study conditions within a single study visit lasting up to 3 hours.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Young Adult EC Users - 20mg/mL, 5% Free-base: Young Adult EC Users - 20mg/mL nicotine concentration, 5% Free-base fraction
- Young Adult EC Users - 20mg/mL, 25% Free-base: Young Adult EC Users - 20mg/mL nicotine concentration, 25% Free-base fraction
- Young Adult EC Users - 20mg/mL, 45% Free-base: Young Adult EC Users - 20mg/mL nicotine concentration, 45% Free-base fraction
- Young Adult EC Users - 20mg/mL, 65% Free-base: Young Adult EC Users - 20mg/mL nicotine concentration, 65% Free-base fraction
- Young Adult EC Users - 20mg/mL, 85% Free-base: Young Adult EC Users - 20mg/mL nicotine concentration, 85% Free-base fraction
- Young Adult EC Users - 50mg/mL, 5% Free-base: Young Adult EC Users - 50mg/mL nicotine concentration, 5% Free-base fraction
- Young Adult EC Users - 50mg/mL, 25% Free-base: Young Adult EC Users - 50mg/mL nicotine concentration, 25% Free-base fraction
- Young Adult EC Users - 50mg/mL, 45% Free-base: Young Adult EC Users - 50mg/mL nicotine concentration, 45% Free-base fraction
- Young Adult EC Users - 50mg/mL, 65% Free-base: Young Adult EC Users - 50mg/mL nicotine concentration, 65% Free-base fraction
- Young Adult EC Users - 50mg/mL, 85% Free-base: Young Adult EC Users - 50mg/mL nicotine concentration, 85% Free-base fraction
- Older Adult Smokers - 20mg/mL, 5% Free-base: Older Adult Smokers - 20mg/mL nicotine concentration, 5% Free-base fraction
- Older Adult Smokers - 20mg/mL, 25% Free-base: Older Adult Smokers - 20mg/mL nicotine concentration, 25% Free-base fraction
- Older Adult Smokers - 20mg/mL, 45% Free-base: Older Adult Smokers - 20mg/mL nicotine concentration, 45% Free-base fraction
- Older Adult Smokers - 20mg/mL, 65% Free-base: Older Adult Smokers - 20mg/mL nicotine concentration, 65% Free-base fraction
- Older Adult Smokers - 20mg/mL, 85% Free-base: Older Adult Smokers - 20mg/mL nicotine concentration, 85% Free-base fraction
- Older Adult Smokers - 50mg/mL, 5% Free-base: Older Adult Smokers - 50mg/mL nicotine concentration, 5% Free-base fraction
- Older Adult Smokers - 50mg/mL, 25% Free-base: Older Adult Smokers - 50mg/mL nicotine concentration, 25% Free-base fraction
- Older Adult Smokers - 50mg/mL, 45% Free-base: Older Adult Smokers - 50mg/mL nicotine concentration, 45% Free-base fraction
- Older Adult Smokers - 50mg/mL, 65% Free-base: Older Adult Smokers - 50mg/mL nicotine concentration, 65% Free-base fraction
- Older Adult Smokers - 50mg/mL, 85% Free-base: Older Adult Smokers - 50mg/mL nicotine concentration, 85% Free-base fraction
Arm/Group | Young Adult EC Users - 20mg/mL, 5% Free-base | Young Adult EC Users - 20mg/mL, 25% Free-base | Young Adult EC Users - 20mg/mL, 45% Free-base | Young Adult EC Users - 20mg/mL, 65% Free-base | Young Adult EC Users - 20mg/mL, 85% Free-base | Young Adult EC Users - 50mg/mL, 5% Free-base | Young Adult EC Users - 50mg/mL, 25% Free-base | Young Adult EC Users - 50mg/mL, 45% Free-base | Young Adult EC Users - 50mg/mL, 65% Free-base | Young Adult EC Users - 50mg/mL, 85% Free-base | Older Adult Smokers - 20mg/mL, 5% Free-base | Older Adult Smokers - 20mg/mL, 25% Free-base | Older Adult Smokers - 20mg/mL, 45% Free-base | Older Adult Smokers - 20mg/mL, 65% Free-base | Older Adult Smokers - 20mg/mL, 85% Free-base | Older Adult Smokers - 50mg/mL, 5% Free-base | Older Adult Smokers - 50mg/mL, 25% Free-base | Older Adult Smokers - 50mg/mL, 45% Free-base | Older Adult Smokers - 50mg/mL, 65% Free-base | Older Adult Smokers - 50mg/mL, 85% Free-base
Number analyzed (Participants) | 66 | 66 | 66 | 66 | 66 | 66 | 66 | 66 | 66 | 66 | 67 | 66 | 66 | 66 | 67 | 66 | 66 | 66 | 66 | 66
score on a scale
  Try Product Again | 3.73 (2.01) | 3.88 (1.93) | 3.91 (1.86) | 3.74 (1.79) | 3.55 (1.93) | 3.74 (1.98) | 2.95 (1.86) | 3.00 (1.74) | 2.35 (1.52) | 1.94 (1.38) | 3.85 (2.06) | 3.70 (1.97) | 3.44 (1.92) | 3.80 (2.04) | 2.88 (1.83) | 3.44 (1.76) | 3.03 (1.93) | 2.74 (1.78) | 2.24 (1.61) | 2.20 (1.64)
  Purchase Product for Regular Use | 2.86 (1.85) | 2.95 (1.80) | 2.98 (1.69) | 2.71 (1.71) | 2.70 (1.77) | 2.64 (1.73) | 2.29 (1.76) | 2.09 (1.38) | 1.64 (1.25) | 1.52 (1.14) | 3.21 (1.94) | 3.06 (1.98) | 3.03 (1.98) | 3.11 (2.04) | 2.42 (1.74) | 2.92 (1.78) | 2.47 (1.73) | 2.15 (1.60) | 1.91 (1.49) | 1.74 (1.33)
  Use Product Regularly | 2.83 (1.81) | 3.12 (1.88) | 3.05 (1.77) | 2.76 (1.70) | 2.77 (1.80) | 2.71 (1.79) | 2.27 (1.71) | 2.03 (1.37) | 1.74 (1.27) | 1.52 (1.27) | 3.09 (2.00) | 3.02 (1.99) | 2.79 (1.90) | 2.97 (2.09) | 2.36 (1.74) | 2.85 (1.76) | 2.44 (1.81) | 2.14 (1.65) | 1.85 (1.37) | 1.76 (1.35)

2. Primary Outcome: Intensity of Sensory Attributes
Description: 5-item self-report measure completed following e-cigarette self-administration, using the general Labeled Magnitude Scale (gLMS). Scores range from 0 (no sensation) to 100 (strongest imaginable) with higher scores indicating a greater sensation intensity.
Time Frame: as for outcome 1
Population: Participants who provided valid responses to the gLMS items; responses were missing in two instances
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Young Adult EC Users - 20mg/mL, 5% Free-base | Young Adult EC Users - 20mg/mL, 25% Free-base | Young Adult EC Users - 20mg/mL, 45% Free-base | Young Adult EC Users - 20mg/mL, 65% Free-base | Young Adult EC Users - 20mg/mL, 85% Free-base | Young Adult EC Users - 50mg/mL, 5% Free-base | Young Adult EC Users - 50mg/mL, 25% Free-base | Young Adult EC Users - 50mg/mL, 45% Free-base | Young Adult EC Users - 50mg/mL, 65% Free-base | Young Adult EC Users - 50mg/mL, 85% Free-base | Older Adult Smokers - 20mg/mL, 5% Free-base | Older Adult Smokers - 20mg/mL, 25% Free-base | Older Adult Smokers - 20mg/mL, 45% Free-base | Older Adult Smokers - 20mg/mL, 65% Free-base | Older Adult Smokers - 20mg/mL, 85% Free-base | Older Adult Smokers - 50mg/mL, 5% Free-base | Older Adult Smokers - 50mg/mL, 25% Free-base | Older Adult Smokers - 50mg/mL, 45% Free-base | Older Adult Smokers - 50mg/mL, 65% Free-base | Older Adult Smokers - 50mg/mL, 85% Free-base
Number analyzed (Participants) | 66 | 66 | 66 | 66 | 66 | 66 | 66 | 66 | 66 | 66 | 67 | 66 | 66 | 66 | 67 | 66 | 66 | 66 | 66 | 66
score on a scale
  Throat Hit | 13.05 (13.09) | 13.03 (11.66) | 16.17 (15.00) | 17.53 (15.83) | 21.29 (16.80) | 19.39 (14.46) | 32.97 (22.04) | 36.20 (24.04) | 45.77 (27.57) | 53.39 (26.26) | 17.07 (18.12) | 21.64 (22.48) | 22.92 (20.61) | 22.03 (19.99) | 29.51 (24.68) | 26.82 (21.12) | 34.73 (23.18) | 41.21 (20.75) | 46.15 (27.85) | 53.74 (25.87)
  Sweetness: number analyzed (Participants) | 66 | 66 | 66 | 66 | 66 | 66 | 66 | 66 | 66 | 66 | 67 | 66 | 66 | 66 | 66 | 66 | 66 | 66 | 66 | 66
  Sweetness | 14.36 (15.12) | 13.32 (12.41) | 13.61 (15.89) | 12.39 (14.18) | 11.58 (12.08) | 12.59 (13.75) | 11.27 (14.62) | 9.32 (9.58) | 7.20 (12.65) | 6.15 (10.36) | 17.60 (18.23) | 19.29 (20.34) | 21.92 (19.89) | 20.29 (17.41) | 13.82 (14.36) | 18.44 (17.53) | 12.74 (13.77) | 14.33 (17.41) | 12.21 (15.75) | 10.65 (14.50)
  Bitterness | 11.50 (13.32) | 10.67 (11.18) | 11.68 (12.35) | 16.02 (19.25) | 15.27 (16.17) | 13.80 (12.33) | 22.35 (20.55) | 25.26 (22.19) | 27.58 (23.64) | 33.41 (27.26) | 10.19 (12.35) | 13.39 (16.61) | 17.09 (21.37) | 12.68 (14.76) | 15.73 (17.58) | 20.70 (25.12) | 22.11 (22.27) | 28.48 (23.89) | 27.88 (25.39) | 31.55 (25.81)
  Smoothness | 29.82 (25.14) | 26.21 (20.86) | 29.73 (23.68) | 23.12 (20.00) | 23.71 (17.35) | 24.74 (21.30) | 19.20 (18.60) | 12.02 (11.86) | 11.09 (12.19) | 7.59 (9.33) | 37.04 (26.57) | 35.79 (25.53) | 33.38 (24.49) | 33.74 (26.38) | 25.22 (23.31) | 27.06 (21.31) | 22.52 (21.38) | 19.44 (21.90) | 20.74 (25.11) | 13.92 (17.78)
  Harshness: number analyzed (Participants) | 66 | 66 | 66 | 65 | 66 | 66 | 66 | 66 | 66 | 66 | 67 | 66 | 66 | 66 | 67 | 66 | 66 | 66 | 66 | 66
  Harshness | 12.48 (13.95) | 13.53 (14.79) | 13.02 (13.84) | 15.48 (19.13) | 18.14 (18.26) | 16.44 (14.75) | 28.70 (21.76) | 40.41 (25.62) | 44.53 (27.66) | 53.26 (29.61) | 14.33 (17.77) | 18.03 (21.83) | 18.76 (22.65) | 18.24 (19.73) | 27.88 (27.77) | 27.03 (24.99) | 36.36 (27.28) | 42.77 (24.66) | 47.42 (29.32) | 52.77 (29.00)

3. Primary Outcome: Degree of Liking or Disliking of Sensations
Description: Self-report measure completed following e-cigarette self-administration, using the Labeled Hedonic Scale (LHS). Scores range from -100 (most disliked imaginable) to 100 (most liked imaginable) with higher scores indicating a greater degree of liking.
Time Frame: as for outcome 1
Population: Participants who provided valid responses to the LHS item, LHS data was missing in 7 instances
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Young Adult EC Users - 20mg/mL, 5% Free-base | Young Adult EC Users - 20mg/mL, 25% Free-base | Young Adult EC Users - 20mg/mL, 45% Free-base | Young Adult EC Users - 20mg/mL, 65% Free-base | Young Adult EC Users - 20mg/mL, 85% Free-base | Young Adult EC Users - 50mg/mL, 5% Free-base | Young Adult EC Users - 50mg/mL, 25% Free-base | Young Adult EC Users - 50mg/mL, 45% Free-base | Young Adult EC Users - 50mg/mL, 65% Free-base | Young Adult EC Users - 50mg/mL, 85% Free-base | Older Adult Smokers - 20mg/mL, 5% Free-base | Older Adult Smokers - 20mg/mL, 25% Free-base | Older Adult Smokers - 20mg/mL, 45% Free-base | Older Adult Smokers - 20mg/mL, 65% Free-base | Older Adult Smokers - 20mg/mL, 85% Free-base | Older Adult Smokers - 50mg/mL, 5% Free-base | Older Adult Smokers - 50mg/mL, 25% Free-base | Older Adult Smokers - 50mg/mL, 45% Free-base | Older Adult Smokers - 50mg/mL, 65% Free-base | Older Adult Smokers - 50mg/mL, 85% Free-base
Number analyzed (Participants) | 65 | 66 | 66 | 66 | 66 | 66 | 66 | 66 | 66 | 66 | 67 | 65 | 66 | 65 | 66 | 65 | 66 | 65 | 65 | 66
score on a scale | 8.34 (31.61) | 5.33 (33.35) | 11.83 (29.47) | 5.42 (25.27) | 0.05 (28.63) | 6.89 (31.31) | -8.82 (37.66) | -15.58 (33.41) | -30.00 (34.31) | -40.92 (33.84) | 13.94 (38.88) | 12.85 (39.92) | 7.98 (39.40) | 11.74 (40.03) | -7.30 (40.18) | 1.88 (40.00) | -9.27 (46.73) | -19.18 (41.19) | -27.18 (41.80) | -36.61 (41.33)

4. Secondary Outcome: Subjective Appeal
Description: 12-item modified Cigarette Evaluation Questionnaire (mCEQ) completed following e-cigarette self-administration to assess subjective responses to the e-cigarettes. The 12-item mCEQ includes five subscales: Smoking Satisfaction, Psychological Reward, Aversion, Enjoyment of Respiratory Tract Sensations, and Craving Reduction, with items rated from 1 (not at all) to 7 (extremely likely). Scores for each subscale are calculated as the mean of the individual item responses or the single item. Higher scores indicate greater intensity on that scale.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Young Adult EC Users - 20mg/mL, 5% Free-base | Young Adult EC Users - 20mg/mL, 25% Free-base | Young Adult EC Users - 20mg/mL, 45% Free-base | Young Adult EC Users - 20mg/mL, 65% Free-base | Young Adult EC Users - 20mg/mL, 85% Free-base | Young Adult EC Users - 50mg/mL, 5% Free-base | Young Adult EC Users - 50mg/mL, 25% Free-base | Young Adult EC Users - 50mg/mL, 45% Free-base | Young Adult EC Users - 50mg/mL, 65% Free-base | Young Adult EC Users - 50mg/mL, 85% Free-base | Older Adult Smokers - 20mg/mL, 5% Free-base | Older Adult Smokers - 20mg/mL, 25% Free-base | Older Adult Smokers - 20mg/mL, 45% Free-base | Older Adult Smokers - 20mg/mL, 65% Free-base | Older Adult Smokers - 20mg/mL, 85% Free-base | Older Adult Smokers - 50mg/mL, 5% Free-base | Older Adult Smokers - 50mg/mL, 25% Free-base | Older Adult Smokers - 50mg/mL, 45% Free-base | Older Adult Smokers - 50mg/mL, 65% Free-base | Older Adult Smokers - 50mg/mL, 85% Free-base
Number analyzed (Participants) | 66 | 66 | 66 | 66 | 66 | 66 | 66 | 66 | 66 | 66 | 67 | 66 | 66 | 66 | 67 | 66 | 66 | 66 | 66 | 66
score on a scale
  Satisfaction | 3.19 (1.63) | 3.21 (1.27) | 3.20 (1.32) | 3.09 (1.23) | 2.88 (1.32) | 3.13 (1.39) | 2.53 (1.30) | 2.36 (1.24) | 1.92 (1.01) | 1.57 (0.74) | 3.48 (1.68) | 3.38 (1.77) | 3.26 (1.61) | 3.40 (1.67) | 2.75 (1.64) | 3.16 (1.47) | 2.71 (1.48) | 2.34 (1.52) | 2.12 (1.32) | 1.96 (1.31)
  Psychological Reward | 2.06 (1.07) | 2.19 (1.08) | 2.27 (1.10) | 2.22 (1.11) | 2.22 (1.16) | 2.30 (1.18) | 2.18 (1.07) | 2.09 (0.99) | 2.12 (1.07) | 1.85 (0.72) | 2.30 (1.32) | 2.37 (1.38) | 2.22 (1.09) | 2.38 (1.28) | 2.00 (1.10) | 2.20 (1.12) | 2.10 (1.05) | 1.97 (1.15) | 1.76 (0.83) | 1.93 (1.09)
  Aversion | 1.30 (0.48) | 1.27 (0.45) | 1.33 (0.55) | 1.27 (0.60) | 1.31 (0.65) | 1.58 (0.88) | 1.53 (0.74) | 1.56 (0.76) | 1.59 (0.80) | 1.68 (0.93) | 1.28 (0.57) | 1.33 (0.70) | 1.33 (0.65) | 1.22 (0.53) | 1.43 (0.84) | 1.48 (0.82) | 1.33 (0.71) | 1.42 (0.75) | 1.55 (0.92) | 1.48 (0.80)
  Enjoyment of Respiratory Tract Sensations | 2.88 (1.55) | 3.15 (1.38) | 3.03 (1.38) | 2.88 (1.27) | 2.85 (1.32) | 2.98 (1.39) | 2.52 (1.45) | 2.30 (1.29) | 1.95 (1.26) | 1.56 (0.98) | 3.31 (1.72) | 3.30 (1.87) | 3.14 (1.73) | 3.26 (1.77) | 2.58 (1.64) | 3.17 (1.71) | 2.62 (1.54) | 2.03 (1.58) | 2.00 (1.39) | 1.86 (1.37)
  Craving Reduction | 2.23 (1.49) | 2.53 (1.61) | 2.68 (1.65) | 2.50 (1.65) | 2.70 (1.61) | 2.92 (1.71) | 2.67 (1.66) | 2.42 (1.55) | 2.26 (1.46) | 2.21 (1.60) | 2.78 (1.54) | 2.91 (1.71) | 2.76 (1.55) | 3.02 (1.53) | 2.67 (1.54) | 3.00 (1.44) | 2.65 (1.55) | 2.44 (1.51) | 2.26 (1.38) | 2.32 (1.37)

ADVERSE EVENTS:
Time Frame: Single study visit, Up to 3 hours
Description: We combined adverse event reporting across arms because no adverse events occurred, making separate reporting by dose level unnecessary.
Arm/Group | Young Adult EC Users | Older Adult Smokers
All-Cause Mortality (participants affected / at risk) | 0/70 | 0/80
Serious Adverse Events (participants affected / at risk) | 0/70 | 0/80
Other Adverse Events (participants affected / at risk) | 0/70 | 0/80

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-01-23): https://cdn.clinicaltrials.gov/large-docs/86/NCT05864586/Prot_SAP_000.pdf